CLINICAL TRIAL: NCT05747495
Title: Formation of a Network of Volunteers in Maneuverd of Cardiopulmonary Resuscitation and the Use of the Automated External Defibrillator (AED) in the Rural Area Through a Virtual Platform.
Brief Title: Online Formation in Cardiopulmonary Resuscitation in a Rural Area.
Acronym: RECADE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SLT008/18/00039
Record Dates: First submitted 2023-02-08; First posted 2023-02-28 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-01

CONDITIONS: Cardiac Arrest
Keywords: Out-of-hospital cardiac arrest; Cardiopulmonary resuscitation; Automated external defibrillators; Emergency medical system services; Primary healthcare; Rural Health services
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants registered in the online training in CPR-AED (Experimental): The online training has been designed according to the Catalan Resuscitation Council (CCR) and the European Resuscitation Council (ERC) guidelines. The aim of this training is to provide theoretical and practical knowledge to respond to aid situations (from unconscious people to drowning, both adults and children), as well as the use of the AED.
  The contents are available at the link [https://register.magnore.com/registre-curs-de-reanimacio-cardiopulmonar-dea/].
  Interventions: Other: Online training in CPR-AED

INTERVENTIONS:
Other: Online training in CPR-AED — The online training has been designed according to the Catalan Resuscitation Council (CCR) and the European Resuscitation Council (ERC) guidelines. The aim of this training is to provide theoretical and practical knowledge to respond to aid situations (from unconscious people to drowning, both adults and children), as well as the use of the AED.
  The contents are available at the link [https://register.magnore.com/registre-curs-de-reanimacio-cardiopulmonar-dea/].

SUMMARY:
Background: Sudden death due to cardiorespiratory arrest has a high mortality and in most cases occurs in out-of-hospital. Cardiopulmonary resuscitation (CPR) initiated immediately by witnesses doubles survival. However, rural areas present different challenges regarding the arrival of emergency services. As a result, the rural population could benefit from basic CPR training programs, in order to improve survival in front of a situation of cardiorespiratory arrest. The aim of this study is to evaluate the effectiveness of the online training in CPR-AED carried out by participants in a rural area of Camp de Tarragona.

Methodology: Quasi-experimental design, consisting of 2 phases: Phase 1) Evaluation of the effectiveness of the online training in CPR-AED knowledge; Phase 2) Evaluation of the effectiveness of the online training in CPR-AED maneuvers in simulation at short- and medium- term.

The main variable is the score difference between the pre- and post-training test (phase 1) and the passing or not (pass/fail) of the simulated test (phase 2). Continuous variables will be compared using the Student's t-test or the U-Man Whitney test (depending on normality). For categorical variables, Pearson's Chi-square test will be used. A multivariate analysis will be performed to determine which factors independently influence the main variable.

Applicability and Relevance: The evaluation of the effectiveness of this course will allow it to be extended to different rural territories of the community, contributing to the expansion of knowledge of CPR-AED maneuvers.

DETAILED DESCRIPTION:
STUDY OBJECTIVES

The main objective of this study is to determine the effectiveness of an online training in CPR and AED carried out by participants from a rural area of Camp de Tarragona.

Secondary objectives: 1) To determine the improvement of the CPR knowledge of the participants after the course; 2) To assess the CPR skills of the participants of the online course through a face-to-face simulation with mannequins in the short (1 month) and medium term (6 months).

STUDY DESIGN AND SETTING

This study consists of a quasi-experimental comunitary intervention study without a control group.The flowchart of the study is detailed in figure 1. It will be carried out in two phases:

* PHASE 1. Evaluation of the effectiveness of the online training in CPR-AED knowledge.
* PHASE 2. Evaluation of the effectiveness of the online training in CPR-AED maneuvers in simulation.

Participants are being recruited by the primary care centers that encompass the rural area of Tarragona.

PARTICIPANT'S SELECTION AND RECRUITMENT

The reference population is the inhabitants of 15 municipalities in the rural area of the interior of Tarragona, which involve the countries of Priorat and Baix Camp Nord, including a total of 10,256 inhabitants.

These towns refer to the primary care team of Les Borges del Camp and Cornudella de Montsant, according to the followed distribution:

* Basic health area of Les Borges: Alforja, Les Borges del Camp, Riudecols, Aleixar, Maspujols, Vilaplana and Arbolí.
* Basic health area of Cornudella de Montsant: Poboleda, Cornudella de Montsant, Ulldemolins, Prades, Capafonts, La Febró, La Morera de Montsant and Escaladei.

During a 3-month period prior to the courses, online training will be disseminated to different population groups including police, firemen, teaching staff, health workers, shopkeepers, pharmacists among others. In addition, the course will be offered from the primary care centers to everybody but insisting to the relatives of people with heart disease. Moreover, alliances will be sought with the municipal councils, and informative posters will be distributed.

PROCEDURES

PHASE 1. Evaluation of the effectiveness of the online training in CPR-AED knowledge.

People interested in participating must register on a Moodle environment platform. First registration steps will consist of a brief questionnaire with the eligibility criteria and informed consent to participate in the study.

Once registered and during one month they have free access to complete the course, which requires a dedication of 3-4 hours. They can access the platform 7 days a week, 24 hours a day.

Enrolled people will complete two questionnaires, one to assess prior knowledge (Pre-training test) and another, acquired knowledge (Post-training test).

The qualification will be pass or fail. All suitable people will obtain a course certificate and will be invited to be assessed in person by staff accredited by the CCR.

Those who complete the training and are eligible for the assessment will be included in phase II.

PHASE 2. Evaluation of the effectiveness of the online training in CPR-AED maneuvers in simulation.

Volunteers who agree to participate will be invited to face-to-face assessment of CPR skills and use of the AED at short term (1 month) and medium term (6 month) after training. The evaluation will be external to the team that designed the course. The participant will be exposed to an CPA situation and will have to solve according to the acquired competence in CPR and use of the AED, to attend to the affected person (in this case simulated). This evaluation will follow the recommendations described by the ERC. At the end, all competent people will obtain a certified accreditation.

SAMPLE SIZE

For phase 1, the online training course is open access, so anyone who meets the study's selection criteria will be able to take part. For phase 2, of all the people who have completed the course in phase 1 of the study, a representative selection will be made of the reference population covering different age and gender ranges. In addition, the population of participants will be selected proportionally to population density.

In order to evaluate the effectiveness of the training in the simulation, the necessary sample has been calculated with the statistical software GRANMO (IMIM, 2012) using the option of averages observed with respect to a reference sample.

Accepting an alpha risk of 0.05 and a beta risk of 0.2 for a bilateral contrast, it is considered that 52 participants are needed to detect a difference equal to or greater than 0.5 points in the face-to-face evaluation of the online training. A common standard deviation of 1.07* is assumed.

The number of subjects is increased by 30% assuming a forecast of losses to follow-up.

DATA COLLECTION

For phase 1, data will be collected through the online training platform and stored in an electronic format on a personal device, under the supervision of the principal investigator. Access is controlled with credentials. The data obtained will be used only for this study for the purpose of the same.

For phase 2, data is collected through the CCR questionnaire (Annex 5) by the health professional with CCR accreditation.

STATISTICAL ANALYSES

Quantitative variables will be expressed as mean (± standard deviation), if they follow a normal distribution, or in median and interquartile range if they do not follow a normal distribution. The normality of the variables will be described using the Kolmogorov test.

Qualitative variables will be described with percentages and 95% confidence intervals. The usual statistical tests will be used in this type of study.

Initially, a descriptive analysis of the study population and a bivariate analysis will be carried out, separating the cohort between the participants who were PASS or NOT PASS the simulation. Finally, a multivariate analysis will be performed to determine which factors independently influence the main variable, adjusting all the variables of interest described above. It will be performed with a linear regression.

ELIGIBILITY:
Inclusion Criteria:

* Residing in the rural area of Priorat and Baix Camp Nord.
* >18 years old
* Having a device with internet connection
* Be interested in taking part in the virtual course as a participants

Exclusion Criteria:

* Language troubles
* Disability that prevents from carrying out the CPR and AED course and measures
* Difficulty attending practical sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the online training in CPR-AED knowledge | 1 month
  The score difference obtained between the pre-training test and the post-training test.
Effectiveness of the online training in CPR-AED maneuvers in simulation | 6 months
  The CCR checklist will be used to evaluate the maneuvers in simulation. This variable will be defined as dichotomous. If the participant's result is APPROVED, he will be considered PASSED and if the result is FAILED, he will be NOT APPROVED.

SECONDARY OUTCOMES:
Socio-demographic data | 1 month
  Age, gender, population of residence, education level, socioeconomic level.
ACP data | 1 month
  Previous training in CPR, family or personal history of heart disease or other risk factors, having previously witnessed an ACP, previous performance before ACP assessed through a questionnaire
Time taken to complete the course | 1 month
  Once registered and during one month participants have free access to complete the course, which requires a dedication of 3-4 hours.
The number of entries to complete the course | 1 month
  Participants can access the platform 7 days a week, 24 hours a day.
Data on the satisfaction questionnaire | 1 month
  Final score (1-5) and by dimensions (organization, methodology, applicability, general assessment, teacher assessment) .

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Rey-Reñones, PhD, Principal Investigator — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Locations (1):
- IDIAP Jordi Gol, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared. Results obtained in the simulation environment will be delivered to the participant himself through email.
  Results will be published by the investigators in academic journals, newapapers and social media.

REFERENCES:
- [Derived] Taverna-Llaurado E, Martinez-Torres S, Granado-Font E, Palleja-Millan M, Del Pozo A, Roca-Biosca A, Martin-Lujan F, Rey-Renones C. Online platform for cardiopulmonary resuscitation and automated external defibrillator training in a rural area: a community clinical trial protocol. BMJ Open. 2024 Feb 7;14(2):e079467. doi: 10.1136/bmjopen-2023-079467. PMID 38326271